CLINICAL TRIAL: NCT04577638
Title: A Phase II Trial Evaluating Conformational Intensity Modulated Radiotherapy With Concomitant Nivolumab Followed by Nivolumab for Patients With Locally Advanced Non-small Cell Lung Cancer
Brief Title: Accelerated Radio-Immunotherapy for Lung Cancer
Acronym: AIRING
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Center Eugene Marquis (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-1-39-007
Record Dates: First submitted 2020-09-30; First posted 2020-10-08 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Non Small Cell Lung Cancer Stage III
Keywords: Immunotherapy; Accelerated Intensity Modulated Radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab and accelerated IMRT (Experimental)
  Interventions: Combination Product: Nivolumab and Intensity Modulated Radiotherapy (IMRT)

INTERVENTIONS:
Combination Product: Nivolumab and Intensity Modulated Radiotherapy (IMRT) — Every included patient will receive the experimental treatment regimen as follows:
  * Combination of IMRT 66 Gray (Gy)/24 fractions of 2.75 Gy) and immunotherapy with 3 doses of nivolumab, 240 mg (1th, 3th and 5th week of IMRT) during 5 weeks
  * Maintenance treatment by nivolumab 240 mg (Q2W) during 6 months, or until progression and severe toxicity leading to definitive treatment interruption.

SUMMARY:
Radiotherapy (RT), at a total dose of 60-66 Gy over 6 weeks, combined with platinum-based chemotherapy, is the standard of care for stage III Non-Small Cell Lung Cancers (NSCLC) patients with unresectable or inoperable disease. However, the long-term outcomes are poor, with a 5-year overall survival (OS) rate of 15-35% for stage IIIA, and 5-10% for stage IIIB patients. The recent association of immunotherapy has been proven to improve Progression Free Survival (PFS) and OS for these patients and durvalumab consolidation following chemoradiotherapy (CT-RT) is now the new standard of care.

Compared to older technics (2Dimensions(D) and 3D-RT), intensity-modulated radiotherapy (IMRT) allows for improved organs-at-risk sparing, owing to the high dose conformation to the target volume, thus reducing toxicity rates.

In regard to the recent results of adjuvant immunotherapy, the benefits of concomitant chemotherapy with radiotherapy could be re-evaluated. With the changing landscape in the standard treatment of Local Advanced NSCLC (LA-NSCLC), the reduction in treatment-induced toxicity, while maintaining optimal tumor control, has become a priority, thereby warranting access to adjuvant immunotherapy for these patients. Due to the toxicity of the chemoradiotherapy, a large subset of patients may be unfit for the adjuvant immunotherapy. The use of immunotherapy concomitant to radiotherapy without chemotherapy may be the next step. Nevertheless, as immune cells are highly sensitive to conventional RT doses, the paradigm of the standard irradiation volumes should be reconsidered. In this context, the introduction of IMRT to spare lymphatic tissues and bone marrow deserves evaluation in prospective trials.

A strong body of evidence supports the combination of RT with immunotherapy such as a Programmed cells Death-1 (PD1) inhibitor. Radiation alone can modify the immune response in several ways to allow for synergistic effects when combined with immunotherapy.

The reduction in treatment-induced toxicity while maintaining optimal tumor control has become a priority, thereby warranting access to adjuvant immunotherapy for these patients. In this context, the introduction of IMRT to spare lymphatic tissues and bone marrow deserves evaluation in prospective trials.

The timing of administration of immunotherapy seems to be a major point. Previous data in mice showed that an improved survival benefit with concurrent anti-PD-Ligand1 (PD-L1) and RT versus sequential administration. Moreover, for sequential schedule, an improved survival outcome was found for patients receiving first dose of durvalumab within 14 days of last radiotherapy fraction compared to 14 days or greater.

Furthermore, immunotherapy combined with radiotherapy appears to be safe, without increase of the toxicity.

In summary, there is a strong rationale for testing this new paradigm of accelerated IMRT combined with concurrent and maintenance nivolumab for locally advanced non-small lung cancer, due to:

* The unmet medical need for new Standard Of Care (SOC) better tolerated and " as " or " more " effective treatment than CT-RT
* The need to decrease radiation-induced toxicity
* The limit of CT-RT followed by durvalumab consolidation, leading to a high rate of recurrence within the 18 months (18-month PFS rate of 44.2%)
* The strong rationale to combine RT and PD-1 inhibition

It is hypothesized this innovative concept to be safe in the context of this study for the following reasons:

* The use of moderate accelerated intensity-modulated radiotherapy (H-IMRT) allows decreasing both the Overall Treatment Time (OTT) and the dose to the organs at risk
* The decrease of the OTT (24 fractions instead of 33 fractions) combined with a decrease of the toxicity should represent a potential clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Stage III non-small lung cancer;
* Patient with at least one of these fragility criteria:

  * Status ECOG 1 with multiple comorbidities, at least 2 pathologies with grade ≥ 2 (renal and/or cardiac and/or vascular and/or hepatic, and/or neurologic, and/or pulmonary)
  * Status ECOG = 2
  * Age > 74 years
  * Age ≥ 70, unfit to receive chemotherapy
* Eligible to radiotherapy, defined by multidisciplinary tumor board;
* Performance Status Eastern Cooperative Oncology Group (ECOG) 0-2;
* Age ≥ 18 years;
* Metastasis (M)0 based on clinical, Magnetic Resonance Imaging (MRI) of brain and FluoroDeoxyGlucose (FDG)/ Positron Emission Tomography (PET)- computerized tomography (CT) examinations;
* Written informed consent

Exclusion Criteria:

* Patients eligible to surgery
* Any prior or current treatment for invasive lung cancer
* History of other malignancy within the last 3 years (exception of in situ carcinoma, skin carcinomas, localized prostate carcinoma Gleason 6 and in situ breast carcinoma)
* Significant disease which, in the judgment of the investigator, as a result of the medical interview, physical examinations, or screening investigations would make the patient inappropriate for entry into the trial
* Known hypersensitivity reaction to nivolumab
* Prior organ transplantation including allogenic stem-cell transplantation
* Any social, personal, medical and/or psychologic factor(s) that could interfere with the observance of the patient to the protocol and/or the follow-up and/or the signature of the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of the efficacy (disease control rate) of accelerated IMRT combined with nivolumab as a first treatment line for patients with a locally advanced non-small cell lung cancer unfit for concomitant or sequential chemoradiotherapy and surgery. | Control of the disease one year after treatment start

CONTACTS AND LOCATIONS:
Overall Officials: Joël Castelli, MD, Principal Investigator — Centre Régional de Lutte Contre le Cancer Eugène Marquis
Locations (5):
- France (5):
  - Centre Hospitalier de Brest, Brest
  - Centre de Lutte Contre le Cancer François Baclesse, Caen
  - Centre de Lutte contre le Cancer Oscar Lambret, Lille
  - Valérie JOLAINE, Rennes
  - Institut de Cancérologie de l'Ouest, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No